CLINICAL TRIAL: NCT04642456
Title: Development and Reliability of a Balance Assessment Scale and Trunk Strength Measurement Protocol to Measure Functionality in Adults With Spinal Deformity
Brief Title: Balance Assessment Scale and Strength Measurement Protocol to Measure Functionality in Adults With Spinal Deformity
Acronym: F-ASD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: S61860
Record Dates: First submitted 2020-11-16; First posted 2020-11-24 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Spinal Deformity
MeSH Terms: interventions — Electromyography

STUDY DESIGN:
Intervention Model Description: control group with healthy subjects and patient group with spinal deformity (ASD)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Other): Healthy subjects or volunteers
  Intervention:
  Balance Assesment Scale Trunk strength measurement with EMG MRI spine/pelvis EOS stereoradiographic full body exam
  Interventions: Diagnostic Test: Balance Assessment Scale; Diagnostic Test: Trunk strength measurement with EMG; Diagnostic Test: MRI spine/pelvis; Diagnostic Test: EOS stereoradiographic full body exam
- ASD group (Other): Patient group with ASD
  Intervention:
  Balance Assesment Scale Trunk strength measurement with EMG MRI spine/pelvis 2 EOS stereoradiographic full body exam Balance Assesment Scale 2 Trunk strength measurement with EMG 2
  Interventions: Diagnostic Test: Balance Assessment Scale; Diagnostic Test: Trunk strength measurement with EMG; Diagnostic Test: MRI spine/pelvis; Diagnostic Test: EOS stereoradiographic full body exam; Diagnostic Test: Balance Assessment Scale 2; Diagnostic Test: Trunk strength measurement with EMG 2

INTERVENTIONS:
Diagnostic Test: Balance Assessment Scale — The newly developed balance, based on the Balance Evaluation Systems Test (BESTest) and Trunk Control Measurement Scale (TCMS), will be administered by two raters (normative and clinical database + interrater reliability)
Diagnostic Test: Trunk strength measurement with EMG — A trunk strength protocol in sitting position, using a hand-held dynamometer is developed. During the trunk strength measurements muscle activity of certain muscles of the trunk will be measured using surface electromyography (EMG)
Diagnostic Test: MRI spine/pelvis — We will be capturing 3D Magnetic Resonance (MR) images of the subject lying supine with extended knees, using a T1 weighted spine-echo (SE) sequence with interslice distance 3 mm in the area of the hip) extended with full spine MRI images (sagittal full spine T1- and T2- weighted images as part of the standard sagittal view of full spine to check for significant stenosis or spinal cord pathology) and additional T1-weighted axial slices at level L4, T12 and T8 with interslice distance 4 mm.The field of view covers the full spine, pelvis and hip smaller trochanter.
Diagnostic Test: EOS stereoradiographic full body exam — Every subject included in the study will undergo a stereoradiographic full body EOS exam completed with Gravity Line (GL) location, recorded by a force plate on the floor
Diagnostic Test: Balance Assessment Scale 2 — Repeating the newly developed balance test (test-retest reliability) within 2 weeks after first measurement
  Arms: ASD group
Diagnostic Test: Trunk strength measurement with EMG 2 — Repeating the trunk strength protocol with EMG within 2 weeks after the first measurement (test-retest reliability)
  Arms: ASD group

SUMMARY:
Develop reliable methods for functional assessment, for both balance and trunk strength, of Adult Spinal Deformity (ASD) patients and create a first clinical and normative database

1. Compare functionality of ASD and control subjects
2. Relate functionality of ASD patients to their pathology, in terms of spinal deformity and muscle condition

DETAILED DESCRIPTION:
The overall aim of the project is to initiate the shift from 2D to 3D mechanically correct and dynamically informed decision-making in Adolescent Idiopathic Scoliosis (AIS), by identifying and integrating the key parameters that overcome the present limitations of 2D static AIS care. Within the timeframe of the project, we will not be able to identify and integrate the key parameters that will overcome all undesired surgical outcomes and therefore, in addition to the overall surgical outcome assessed by patient reported outcome measures (PROMs) we will specifically focus on post-surgery shoulder balance. Since an elevated shoulder after surgery is one of the most common undesired surgical outcomes (approximately 16% of the treated AIS patients) linked with treatment satisfaction and psychological well-being.

To achieve the overall aim, the project comprises two objectives that will allow us to advance towards 3D dynamically informed decision-making in AIS care:

1. To shift towards a 3D mechanically correct overview of the spinal deformity. The current state-of-the-art guidelines for the selection of fusion levels in AIS patients are based on 2D static radiographic parameters[26]. In order to improve the current state-of-the-art evaluation method, efforts should be made towards a 3D dynamic visualization of the deformity, especially considering that AIS is a 3D deformity of the spine. In addition, the treating surgeon has only limited information on the mechanical behavior of the spine of the AIS patient as the traction radiograph tests that show the displacement of the spine are typically only assessed qualitatively. To overcome this issue, the spine stiffness should be incorporated in order to thrive towards a biomechanically-informed state-of-the-art 3D model.
2. To identify the key 3D parameters that should be considered by the surgeon Once a biomechanically-informed subject specific 3D model that incorporates the mechanical behavior of the spine is developed within objective 1, the crucial next step will be to identify the key parameters that have the potential to improve the clinical decision-making in AIS. As highlighted before, we will focus on post-surgery shoulder balance and the PROMs.

ELIGIBILITY:
Inclusion criteria pathological subjects:

1. Adult (>18 years old) subjects suffering from a adult spinal deformity with sagittal or coronal plane misalignment diagnosed on EOS imaging.
2. Ability to walk at least 50 meters distance independently without a walking aid.
3. No documented neurological disease or vestibular lesion affecting balance nor a current history of musculoskeletal disorders of the lower extremities affecting motor performance.

Inclusion criteria control group:

1. Adults (> 18 year old)
2. No current history of back pain and spinal deformity.
3. Ability to walk at least 1000 meters distance independently without a walking aid.
4. No documented neurological disease or vestibular lesion affecting balance nor a current history of musculoskeletal disorders of the lower extremities affecting motor performance.

Exclusion criteria ASD patients:

1. Age < 18 years old and > 79 years old
2. Absence of adult spinal deformity
3. Non-ability to walk at least 50 meters distance independently, with or without a walking aid.
4. Missing patient informed consent
5. Patients presenting with a neurological disease affecting balance other than Parkinson's disease such as stroke and/or Vestibular lesion
6. Patients with a history of spinal fusion surgery.
7. Patients with a current history of diagnosed musculoskeletal disorders of the trunk and/or lower extremities affecting the motor performance such as severe hip arthrosis with or without flexion contracture, severe knee arthrosis, severe ankle arthrosis, severe leg length discrepancy (> 3 cm)

Exclusion criteria control group:

1. Age < 18 years old and > 79 years old
2. Backpain and/or Sciatica at time of the study
3. Presence of adult spinal deformity leading to a pathological sagittal alignment
4. Non-ability to walk at least 1000 meters distance independently without a walking aid
5. Missing patient informed consent
6. Patients presenting with a neurological disease affecting balance such as Stroke, Parkinson's disease and/or Vestibular lesion
7. Patients with a current history of diagnosed musculoskeletal disorders of the trunk and/or lower extremities affecting the motor performance such as severe hip arthrosis with or without flexion contracture, severe knee arthrosis, severe ankle arthrosis, severe leg length discrepancy (> 3 cm)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Balance performance on the newly developed ASD specific balance scale | Day 1
  Balance performance is measured by two raters to assess interrater reliability of the new scale. Patients will also return within two weeks after the first measurement and repeat the balance assessment to assess the test-retest reliability. Data on both ASD patients and Controls will also serve as a first normative and clinical database.
Balance performance on the newly developed ASD specific balance scale | Day 2
  Balance performance is measured by two raters to assess interrater reliability of the new scale. Patients will also return within two weeks after the first measurement and repeat the balance assessment to assess the test-retest reliability. Data on both ASD patients and Controls will also serve as a first normative and clinical database.
Trunk muscle strength | Day 1
  Trunk muscle strength is measured with a hand-held dynamometer and repeated within two weeks after the first measurement to assess test-retest reliability.Data of ASD patients and controls will also serve as a first normative and clinical database.
Trunk muscle strength | Day 2
  Trunk muscle strength is measured with a hand-held dynamometer and repeated within two weeks after the first measurement to assess test-retest reliability.Data of ASD patients and controls will also serve as a first normative and clinical database.

SECONDARY OUTCOMES:
Echointensity of trunk muscles on MRI | Day 1
  Fatty infiltration of trunk muscles is measured by the difference in echointensity on MRI images. This will be related to balance performance and trunk muscle strength.
Static 2D radiographic evaluation of spinopelvic parameters | Day 1
  Spinopelvic parameters are obtained on biplanar radiographic images. These will be related to balance performance and trunk muscle strength.

CONTACTS AND LOCATIONS:
Overall Officials: Lieven Moke, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium